CLINICAL TRIAL: NCT00295854
Title: A Phase II, Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate the Efficacy and Safety of Two Dosing Regimens of MN-001 in Patients With Interstitial Cystitis
Brief Title: Phase II Study Efficacy and Safety of Two Dosing Regimens of MN-001 in Patients With Interstitial Cystitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MN-001-CL-002
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Results first posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-12

CONDITIONS: Interstitial Cystitis
Keywords: Interstitial Cystitis; urgency; frequency; MN-001; Global Response Assessment; bladder pain/urgency; O'Leary Sant IC Symptom and Problem Index
MeSH Terms: conditions — Cystitis, Interstitial | interventions — 4-(6-acetyl-3-(3-(4-acetyl-3-hydroxy-2-propylphenylthio)propoxy)-2-propylphenoxy)butyric acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MN-001 (Experimental)
  Interventions: Drug: MN-001 BID; Drug: MN-001
- MN-001 once daily (Placebo Comparator): placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MN-001 BID — Eligible patients received 500 mg MN-001 bid
  Arms: MN-001
Drug: MN-001 — Eligible patients received 500 mg MN-001 once daily (qd)
  Arms: MN-001
Drug: Placebo — Eligible patients received placebo
  Arms: MN-001 once daily

SUMMARY:
To evaluate the safety and efficacy of 8 weeks of treatment with MN-001 at 500 mg bid, 500 mg once daily vs. placebo in patients with Interstitial Cystitis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-center study to evaluate the efficacy and safety of two dosing regimens of MN-001 in patients with Interstitial Cystitis (IC). Patients will be screened for study eligibility within seven to nine days of randomization. Eligible patients will be randomized in a 1:1:1 ratio to receive either 500 mg MN-001 bid, 500 mg MN-001 once daily or placebo. Patients will be dispensed study drug beginning at Baseline (Visit 2) and will return to the study center for Visit 3 (28 days ± 2 days after Baseline), and Visit 4 (56 days ± 2 days after Baseline), at end of study for safety and efficacy assessments. The patient will be contacted by telephone at Week 6 (42 days ± 2 days after Baseline) for an interim follow up. Study drug will be dispensed at Visits 2 and 3. Safety assessments will include adverse events, physical examinations, clinical laboratory testing, and changes in vital signs. Efficacy assessments include percentage of patients at least "moderately improved" for each treatment group using the patient reported Global Response Assessment (GRA) (see Appendix 1). Secondary assessments include a decrease in bladder pain/urgency based on change in the patient rating from baseline to endpoint using the GRA (see Appendix 1), modified Pelvic Pain and Urgency/Frequency (PUF) Patient Symptom Scale (see Appendix 2) and the O'Leary Sant IC Symptom and Problem Index.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age with a diagnosis of moderate to severe IC;
* Bladder pain ≥ 6 months prior to baseline;
* Urinary frequency of ≥ 8 ≤ 30 micturitions within 24 hours while awake;
* Nocturia ≥ 2x/night;
* Males and females of child-bearing potential (not surgically sterile or post-menopausal) must be abstinent or agree to use an study-accepted contraceptive regimens throughout the study:
* Female patients of child bearing age must have a negative urine pregnancy test at screening;
* Must provide a signed informed consent.

Exclusion Criteria:

* Male or females < 18 years of age;
* Initiation of new IC medication ≤ 30 days prior to baseline;
* Treatment with Elmiron ≤ 120 days prior to baseline;
* Treatment with bladder hydro-distention ≤ 6 months prior to baseline;
* Treatment with intravesical therapy ≤ 60 days prior to baseline;
* History of previous procedure(s) (e.g., augmentation cytoplasty, cystectomy or cystolysis) that has affected bladder function;
* Active genital herpes or vaginitis ≤ 90 days prior to baseline;
* Urinary tract or prostatic infection ≤ 90 days prior to baseline;
* History of urethral diverticulum;
* History of bladder or ureteral calculi;
* History of cyclophosphamide or chemical cystitis, urinary tuberculosis or radiation cystitis;
* History of bladder tumors;
* History of uterine, cervical, vaginal, prostatic or urethral cancer ≤ 5 years prior to baseline;
* Patient is currently pregnant, lactating or likely to become pregnant during the study;
* Participated in another clinical study with an investigational drug or device ≤ 30 days prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2005-05; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Gammans, MD, Study Director — MediciNova, Inc.
Locations (28):
- United States (28):
  - MediciNova Investigational Site, Birmingham, Alabama
  - Citrus Valley Urological Medical Group, Glendora, California
  - Atlantic Urological Medical Group, Long Beach, California
  - Mendez Transplant and Urological Medical Group, San Diego, California
  - Boulder Medical Center, P.C., Boulder, Colorado
  - Western Urologic Research Center, Wheat Ridge, Colorado
  - Segal Institute for Clinical Research, Aventura, Florida
  - Visions Clinical Research, Boynton Beach, Florida
  - West Florida Urology, Palm Harbor, Florida
  - Adult and Pediatric Urology, Plantation, Florida
  - Georgis Patsias, MD., PA, Wellington, Florida
  - Shepherd Center, Inc., Atlanta, Georgia
  - Center For Advanced Pelvic Surgery, Centralia, Illinois
  - Evanston Continence Center, Evanston, Illinois
  - Regional Urology, LLC, Shreveport, Louisiana
  - William Beaumont Hospital, Royal Oak, Michigan
  - Sheldon J. Freedman, MD, LTD, Las Vegas, Nevada
  - Associated Urologic Specialists, P.A., Marlton, New Jersey
  - Upstate Urology, Albany, New York
  - Lyndhurst Gynecology Associates, Winston-Salem, North Carolina
  - Tristate Urologic Services PSC., Inc., Cincinnati, Ohio
  - Midwest Regional Center For Chronic Pelvic Pain and Bladder Control, Lima, Ohio
  - Williamette Women's Healthcare P.C., Tualatin, Oregon
  - The Urology Group, Greer, South Carolina
  - Medical Arts Clinic, Corsicana, Texas
  - Gant Foundation, Fort Worth, Texas
  - Brian Heaton, MD, Ogden, Utah
  - Integrity Medical Research, LLC, Mountlake Terrace, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for study eligibility within 7-9 days of randomization. Patients underwent screening at Visit 1 (≤ 7 days prior to Baseline) and additional eligibility assessments prior to randomization at Visit 2 (Baseline Visit, Day 0).
Pre-assignment Details: Eligible patients were randomized in a 1:1:1 ratio to receive 500 mg MN-001 twice daily (BID), 500 mg MN-001 once daily (QD), or placebo. Patients returned to the study center at Visit 3 (Day 28) and at Visit 4 (Week 8, Day 64) for safety and efficacy assessments. Patients were dispensed study drug at Baseline (Visit 2) and Visit 3.
Groups:
- MN-001 500 mg qd: This group received MN-001 500mg orally (PO)once a day. Patients underwent screening at Visit 1 (≤ 7 days prior to Baseline) and additional eligibility assessments at Visit 2 (Baseline Visit) prior to randomization and after randomization, were scheduled to return at Visit 3 (28 days ± 2 days after Baseline) and at Visit 4 (Week 8, 64 ± 2 days after Baseline) for safety and efficacy assessments. Patients were dispensed study drug at Baseline (Visit 2) and Visit 3. The patients were contacted by telephone at Week 6 (42 days ± 2 days after Baseline) for an interim follow up.
- MN-001 500 mg BID: Patients received MN-001 500 mg BID. Patients underwent screening at Visit 1 (≤ 7 days prior to Baseline) and additional eligibility assessments at Visit 2 (Baseline Visit) prior to randomization and after randomization, were scheduled to return at Visit 3 (28 days ± 2 days after Baseline) and at Visit 4 (Week 8, 64 ± 2 days after Baseline) for safety and efficacy assessments. Patients were dispensed study drug at Baseline (Visit 2) and Visit 3. The patients were contacted by telephone at Week 6 (42 days ± 2 days after Baseline) for an interim follow up.
- Placebo: Patients received placebo. Patients underwent screening at Visit 1 (≤ 7 days prior to Baseline) and additional eligibility assessments at Visit 2 (Baseline Visit) prior to randomization and after randomization, were scheduled to return at Visit 3 (28 days ± 2 days after Baseline) and at Visit 4 (Week 8, 64 ± 2 days after Baseline) for safety and efficacy assessments. Patients were dispensed study drug at Baseline (Visit 2) and Visit 3. The patients were contacted by telephone at Week 6 (42 days ± 2 days after Baseline) for an interim follow up.
Period: Overall Study
Arm/Group | MN-001 500 mg qd | MN-001 500 mg BID | Placebo
Started | 95 | 108 | 102
Safety Population (N=304) | 95 | 108 | 101
ITT Population (N=296) | 92 | 105 | 99
Completed | 77 | 87 | 87
Not Completed | 18 | 21 | 15
Not completed — Adverse Event | 7 | 7 | 6
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 7 | 4
Not completed — did not continue to meet criteria | 1 | 1 | 2
Not completed — required a prohibited medication | 1 | 0 | 0
Not completed — Other | 3 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MN-001 500 mg qd | MN-001 500 mg BID | Placebo | Total
Number analyzed (Participants) | 95 | 108 | 102 | 305
Age Continuous [Mean (Standard Deviation); unit: years] | 45.2 (12.87) | 43.5 (13.95) | 43.4 (13.97) | 44 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 97 | 92 | 271
  Male | 13 | 11 | 10 | 34
Region of Enrollment [Number; unit: participants]
  United States | 95 | 108 | 102 | 305
diagnosis of moderate to severe interstitial cystitis (IC) with bladder pain for ≥ 6 months [Number; unit: participants] — Diagnosis of moderate to severe interstitial cystitis (IC) with bladder pain for ≥ 6 months prior to Baseline, a score of ≥ 15 on the Modified Pelvic Pain and Urgency/Frequency (PUF) Patient Symptom Scale, a score of ≥ 12 on the O'Leary Sant IC Symptom and Problem Index, urinary frequency of ≥ 8 ≤ 30 micturitions within 24 hours while awake, and a history of nocturia ≥ 2 x/night over an 8-hour period prior to screening or Baseline.
  participants
    <=18 years | 0 | 0 | 0 | 0
    Over 18 years old | 95 | 108 | 102 | 305

OUTCOME MEASURES:

1. Secondary Outcome: Number of Responders for GRA Assessment in Their Condition at Week 4.
Description: Responders were defined as patients who were 'moderately improved' or 'markedly improved' and non-responders were defined as patients who were 'markedly worse', 'moderately worse', 'mildly worse', no change, or 'mildly improved' on the GRA assessments.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | MN-001 500 mg qd | MN-001 500 mg BID | Placebo
Number analyzed (Participants) | 92 | 105 | 99
participants | 19 | 26 | 12

2. Primary Outcome: Number Subjects at Least "Moderately Improved" for Each Treatment Group in Patient Reported Global Response Assessment (GRA)
Description: The primary endpoint was the GRA overall change "in their condition" at Week 8. Each patient completed the questionnaire that rated the improvement in their IC symptoms based on responses to the GRA questions. Each question asked the patient to describe the OVERALL CHANGE in pain, urgency, frequency or overall change in their problem compared to the status before taking the study medication. Each parameter was rated on a 7 point scale: markedly worse, moderately worse, mildly worse, same, mildly improved, moderately improved and markedly improved.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | MN-001 500 mg qd | MN-001 500 mg BID | Placebo
Number analyzed (Participants) | 95 | 108 | 102
participants | 31 | 26 | 30

ADVERSE EVENTS:
Time Frame: The mean days of exposure to study drug was similar in the three treatment groups and ranged between 1 to 69 days. Adverse event reporting started on Day 1 of study drug exposure for each patient who received study drug or placebo.
Description: Safety assessments included adverse events (AEs), physical examinations, vital signs, 12 lead ECGs and clinical laboratory testing.
Arm/Group | MN-001 500 mg qd | MN-001 500 mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 1/92 | 0/105 | 1/99
Other Adverse Events (participants affected / at risk) | 48/92 | 65/105 | 28/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MN-001 500 mg qd (N=92) | MN-001 500 mg BID (N=105) | Placebo (N=99)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) — 22 y.o. patient notified site of pregnancy.Female infant reported to have a severe coloboma of retina, iris.Event was continuing at the time of report.No further information available. P.I. opinion: event was possibly related to the study medication.
infected epidermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — 56 y.o. female,epidermal cyst of R thigh,incision,drainage.Hospitalized for worsening cellulitis and had repeat incision,drainage,excision of the cyst, treated with ABs. Recovered from SAE 2 mo later.TEAE considered possibly related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MN-001 500 mg qd (N=92) | MN-001 500 mg BID (N=105) | Placebo (N=99)
Diarrhea (Gastrointestinal disorders) | 11 (12) | 24 (30) | 5 (5)
Nausea (Gastrointestinal disorders) | 10 (12) | 11 (13) | 7 (7)
Loose stools (Gastrointestinal disorders) | 5 (6) | 14 (16) | 3 (4)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 6 (8) | 3 (3)
Headache (Nervous system disorders) | 9 (10) | 9 (10) | 4 (4)
Dizziness (Nervous system disorders) | 6 (7) | 1 (1) | 2 (2)
Interstitial Cystitis (Renal and urinary disorders) | 5 (5) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less